## Dosing strategies for de novo once-daily extended release tacrolimus (LCPT) in kidney transplant recipients

NCT Number: 03713645

**Date: August 21, 2018** 

Descriptive statistics were used to characterize the baseline demographics of the entire cohort (intent to treat population). Continuous parametric data are presented as mean  $\pm$  standard deviation while continuous non-parametric data are presented as median (25%-75% interquartile range). Analysis of outcomes according to CYP3A5 expresser status within the modified ITT population were completed using the Kruskal-Wallis or ANOVA test for continuous data and the chi-squared test for categorical data. Tests were corrected for multiple comparisons as necessary utilizing the Bonferroni method. All tests were two-tailed, and p < 0.05 was used to represent statistical significance. Time to therapeutic tacrolimus trough concentration was analyzed using a Kaplan-Meier time-to-event analysis. All analyses were performed using SPSS, version 26 for windows (Armonk, NY; IBM Inc.).